CLINICAL TRIAL: NCT06443242
Title: Efficacy and Safety of Low-dose Laser Acupuncture on Treating Insomnia Associated With Major Depressive Disorder: A Randomised Controlled Trial
Brief Title: Efficacy and Safety of Low-dose Laser Acupuncture on Treating Insomnia Associated With Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Farris Iman Leong Bin Abdullah (Other)
Collaborators: Henan Medical University (Other)
Responsible Party: Sponsor-Investigator, Mohammad Farris Iman Leong Bin Abdullah, Principal investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XYEFYLL-(Research)-2024-36
Record Dates: First submitted 2024-05-13; First posted 2024-06-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Insomnia
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-Dose Laser Acupuncture (LLA) Group (Experimental): In the Low-Dose Laser Acupuncture (LLA) group, participants receive treatments using the xS-998D06 semiconductor laser acupoint therapeutic device from Nanjing Xiaosong Medical Instruments. This device operates at a wavelength of 780 nm and an output power of 5 mW. Each 20-minute session involves securing the device's probe to specific acupoints (Baihui, Yintang, Anmian, Shenmen, Neiguan, Sanyinjiao, and Taichong) using medical tape. Treatments occur daily for 5 consecutive days each week, with a two-day break, over a 6-week period. All participants, regardless of group assignment, will maintain their regular antidepressant regimen (patients with only one type of antidepressant, such as selective serotonin reuptake inhibitor [SSRI] or serotonin noradrenaline reuptake inhibitor [SNRI] or mirtazapine).
  Interventions: Device: Low-Dose Laser Acupuncture (LLA)
- Sham Laser Acupuncture (SLA) Group (Sham Comparator): Participants in the Sham Laser Acupuncture (SLA) group undergo a sham treatment involving the same procedure and acupoint targeting as the LLA group. The difference lies in the instrument probe being fixed to the acupoint but emitting a dummy laser, simulating the acupuncture experience without actual laser emission. All participants, regardless of group assignment, will maintain their regular antidepressant regimen (patients with only one type of antidepressant, such as selective serotonin reuptake inhibitor [SSRI] or serotonin noradrenaline reuptake inhibitor [SNRI] or mirtazapine).
  Interventions: Device: Sham Laser Acupuncture (SLA)
- Control Group (No Intervention): The control group, which serves as a non-intervention comparison, will continue their standard treatment regimen (patients with only one type of antidepressant, such as selective serotonin reuptake inhibitor [SSRI] or serotonin noradrenaline reuptake inhibitor [SNRI] or mirtazapine).

INTERVENTIONS:
Device: Low-Dose Laser Acupuncture (LLA) — The intervention utilizes the xS-998D06 semiconductor laser acupoint therapeutic device specifically designed for targeted acupoint therapy. This device is critical in delivering precise low-dose laser therapy at a controlled wavelength and power. The laser treatment is directed towards enhancing neurological function and potentially alleviating symptoms of insomnia and depression by stimulating specific acupoints associated with mental health and sleep.
  Arms: Low-Dose Laser Acupuncture (LLA) Group
Device: Sham Laser Acupuncture (SLA) — Sham laser acupuncture serves as a control to assess the placebo effect of the laser treatment. It involves the same procedure as LLA but uses a non-emitting laser probe. This intervention is designed to mimic the LLA setup without delivering actual laser therapy, allowing for an evaluation of the psychological and physiological effects of the placebo compared to the active laser treatment.
  Arms: Sham Laser Acupuncture (SLA) Group

SUMMARY:
The goal of this randomized controlled trial is to assess the efficacy and safety of low-dose laser acupuncture (LLA) in alleviating insomnia symptoms among patients suffering from major depressive disorder.

The study seeks to answer the following questions:

1. How effective is LLA in alleviating insomnia symptoms as compare with SLA and control subjects among patients with major depressive disorder across pre-treatment, mid-treatment and post-treatment assessment?
2. How effective is LLA in alleviating depression symptoms as compare with SLA and control subjects among patients with major depressive disorder across pre-treatment, post-treatment and follow-up assessment?
3. What role do CORT and 5-HT play in the co-occurrence and progression of insomnia and major depressive disorder, and how does LLA act on these mechanisms to provide relief?
4. How does the safety and acceptability of LLA compare to traditional acupuncture in terms of eliminating discomfort and potential side effects? Researchers will compare the effects of LLA with sham laser acupuncture (SLA) and standard medication treatments to evaluate its efficacy and safety.

Participants involved in this study will:

Undergo 30 treatment sessions with LLA or SLA, five times a week for six weeks. Continue their usual pharmacological treatments for major depressive disorder. Participants will undergo comprehensive assessments at key points: pre-treatment, immediately post-treatment, and 12 weeks post-treatment. These evaluations will measure sleep quality and severity of insomnia indices, levels of depression and anxiety, and blood levels of CORT and 5-HT to assess the impact of LLA on insomnia symptoms and biochemical markers. Additionally, participant acceptance and the safety of the treatment will be monitored, including recording any adverse events and medication usage, to determine the effectiveness and safety of LLA in treating insomnia associated with major depressive disorder.

By focusing on these elements, the study aims to provide clear, actionable insights into the benefits and risks of LLA as a treatment option for insomnia associated with major depressive disorder, enhancing the current treatment landscape and patient outcomes.

DETAILED DESCRIPTION:
This randomised controlled trial aims to explore the therapeutic potential of low-dose laser acupuncture (LLA) for treating insomnia in patients diagnosed with major depressive disorder. The study will investigate the physiological and psychological impacts of LLA in comparison with sham laser acupuncture (SLA) and standard pharmacological therapies.

Intervention Details:

LLA involves the application of a low-level laser to specific acupoints known to affect sleep and mood regulation. The technique mimics traditional acupuncture but uses laser light to stimulate these points without physical penetration of the skin, offering a non-invasive alternative with potentially fewer adverse effects. The primary acupoints targeted in this study include Baihui (GV20), Yintang (GV29), Anmian (EX-HN22), Shenmen (HT7), Neiguan (PC6), Sanyinjiao (SP6), and Taichong (LR3).

Study Phases:

The study will be structured into three key phases: pre-treatment, immediately post-treatment, and 12 weeks post-treatment. During the pre-treatment phase, baseline evaluations will be conducted to establish initial levels of insomnia and depressive symptoms in participants. The treatment phase will follow, lasting six weeks, with participants receiving five sessions per week. Subsequent assessments will occur immediately post-treatment to evaluate the immediate effects of the interventions, and again at 12 weeks post-treatment to assess the long-term outcomes.

Research Focus:

The study will particularly focus on the effectiveness of LLA in improving sleep quality as measured by validated scales and objective assessments like actigraphy, which monitors sleep-wake patterns. Additionally, the research will assess changes in psychological state and biochemical markers, which are critical in understanding the interaction between sleep disorders and depression. These measures will help ascertain whether LLA can alter the physiological pathways typically disrupted in major depressive disorder, potentially offering a new avenue for treatment that could complement or reduce the need for pharmacological intervention.

Innovation and Potential Impact:

By integrating a novel, non-invasive method such as LLA, the study could significantly impact the treatment strategies for insomnia in the context of major depressive disorder. This approach not only aims to reduce symptoms but also to enhance overall treatment tolerance and patient adherence, addressing key challenges in managing these interlinked conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients with a diagnosis of major depressive disorder (diagnosed according to the relevant diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders-V).
2. Male or female, 18 to 60 years of age.
3. Participants complaining of insomnia at initial screening.
4. PSQI score over 7.
5. HAMD score between 20 and 35.
6. No use of hypnotic medication or acupuncture treatment within the last month.
7. No cognitive or communication disorders.
8. Willingness to accept random group assignment and sign an informed consent form.
9. Those who have been on stable dose of antidepressant for at least the most recent two weeks and willing to maintain on the same dosage throughout the study.

Exclusion Criteria:

1. Individuals with a marked tendency towards suicide, as assessed by a specialist;
2. Individuals previously diagnosed with schizophrenia, bipolar disorder, or other psychiatric disorders;
3. Individuals with severe alcohol or drug abuse issues;
4. Individuals with liver or kidney dysfunction, or with uncontrollable tumors or significant cerebrovascular diseases;
5. Women who are pregnant or breastfeeding;
6. Individuals likely to have poor compliance or who are fearful of acupuncture treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality from pre-treatment assessed by the Pittsburgh Sleep Quality Index (PSQI) score at immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment.
  This outcome measure evaluates the change in sleep quality in patients with major depressive disorder (MDD) and insomnia treated with Low-Dose Laser Acupuncture (LLA). The Pittsburgh Sleep Quality Index (PSQI) is used, with scores ranging from 0 to 21, where higher scores indicate poorer sleep quality.

SECONDARY OUTCOMES:
Changes in severity of depressive symptoms from pre-treatment assessed by Hamilton Depression Rating Scale (HAMD) score at immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment.
  This outcome measure evaluates the impact of LLA on the severity of depressive symptoms in patients with MDD and insomnia. The Hamilton Depression Rating Scale (HAMD) is used, with scores ranging from 0 to 52, where higher scores indicate more severe depression symptoms.
Changes in severity of insomnia from pre-treatment measure by Insomnia Severity Index (ISI) score at immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment
  This outcome measure assesses the impact of LLA on the change in severity of insomnia in patients with MDD and insomnia across time. The Insomnia Severity Index is used, with scores ranging from 0 to 28, where higher scores indicate more severe degree of insomnia.
Changes in serum corticosterone levels from pre-treatment measure by Immunoassays at immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment.
  This outcome measure examines the change in serum corticosterone levels in patients with MDD and insomnia treated with LLA. Corticosterone levels are measured in ng/mL, with higher levels typically associated with higher stress and worse outcomes.
Changes in serum 5-Hydroxytryptamine (5-HT) levels from pre-treatment measure with Enzyme-Linked Immunosorbent Assay at immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment.
  This outcome measure examines the change in serum 5-hydroxytryptamine (5-HT) levels in patients with MDD and insomnia treated with LLA. 5-HT levels are measured in ng/mL, with lower levels typically associated with worse outcomes in depression and insomnia.
Changes in the incidence of treatment-emergent adverse events from pre-treatment assess as dropout rates at immediately post-treatment and 12 weeks post-treatment | Throughout the study duration (Pre-treatment through 12 weeks post-intervention)
  This outcome measure assesses the incidence of treatment-emergent adverse events to determine the safety of LLA. It compares the dropout rates due to adverse effects among patients in the LLA, Sham Laser Acupuncture (SLA), and control groups.
Changes in the objective sleep patterns (total sleep time, sleep efficacy and number of awakenings) from pre-treatment assess by actigraphy to immediately post-treatment and 12 weeks post-treatment | Pre-treatment, immediately post-treatment and 12 weeks post-treatment
  Description: This outcome measure evaluates the change in objective sleep patterns in patients with MDD and insomnia treated with LLA. Actigraphy provides data on sleep parameters such as total sleep time, sleep efficiency, and number of awakenings.
Monitoring of drug dose record (medication dosage and daily administration time) for any changes from pre-treatment and throughout the 12-week follow-up period of the study | Throughout the study duration (Pre-treatment through 12 weeks post-intervention)
  The dose diary is a record book in which participants will record the medication name, dosage, and exact administration time daily from baseline from pre-treatment through the 12-week follow-up period of the study.
Monitoring of participant compliance to the intervention in the LLA and SLA groups from pre-treatment through the 12-week post-treatment follow-up | Throughout the study duration (Pre-treatment through 12 weeks post-intervention)
  Participants' adherence to the intervention will be recorded in detail. For treatment absences, drop-outs, and loss to follow-up, the causes of non-compliance (such as reduced participation, aversion to the intervention, physical discomfort) will also be documented to ensure integrity and rigor throughout the study.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data will be made available after publication of the study's findings. The data will be uploaded in Figshare data repository after completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be uploaded in Figshare data repository after completion of the study and it will be available for 2 years after completion of the study.
Access Criteria: All researchers and study participants upon request after completion of the study.

REFERENCES:
- [Derived] Qiu Q, Yam MF, Yang W, Guo F, Liu C, Leong Bin Abdullah MFI, Yang S. Efficacy and safety of laser acupuncture for treating insomnia in major depressive disorder: study protocol for a randomized controlled trial. Front Psychiatry. 2025 Nov 20;16:1698773. doi: 10.3389/fpsyt.2025.1698773. eCollection 2025. PMID 41356687